CLINICAL TRIAL: NCT05688176
Title: Liquid Biopsies in Esophageal Adenocarcinoma: Barrett's Esophagus and Esophageal Adenocarcinoma, Searching for Reliable Diagnostic RNA Plasma-based Biomarkers
Brief Title: Barrett's Esophagus and Esophageal Adenocarcinoma, Searching for Reliable Diagnostic RNA Plasma-based Biomarkers
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: B670201628319
Record Dates: First submitted 2018-07-12; First posted 2023-01-18 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms; Liquid biopsy; Transcriptome
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and tissue collection

SUMMARY:
This study is designed to perform a explorative search of the transcriptome to detect new circulating diagnostic sensitive and specific biomarkers in patients with Barrett's esophagus or esophageal adenocarcinoma.

DETAILED DESCRIPTION:
By developing new tools for risk-assessing of Barrett's esophagus (BE) and esophageal adenocarcinoma (EAC) in a population at risk, the investigators expect that diagnosis can be done in an earlier stage resulting in an improved 5-year survival. A proof-of-concept RNA profiling study will be done in 20 BE and EAC patients where 2 biomaterials (tissue and plasma) and 2 RNA biotopes (micro RNA and messenger RNA) will be compared. Previously validated methodology on small RNA and messenger RNA capture sequencing on both tissue and plasma will be used to obtain high-quality data. Differential expression analysis will be done on tissue and plasma sample data. Additional in-depth data-mining will be done, amongst other focusing on structural information encoded in the transcriptome and building a multifeature classifier. These findings will be validated in a large validation cohort, followed by development of a clinical-grade quantitative Polymerase Chain Reaction (qPCR) test, ready for testing in an independent cohort.

ELIGIBILITY:
Inclusion Criteria:

* Barrett's Esophagus with length > 3cm OR esophageal adenocarcinoma histologically proven
* Adequate mental faculty, allowing to understand the proposed treatment protocol and provide informed consent
* Age over 18 years
* No other concurrent malignant disease
* No inclusion in other clinical trials interfering with the study protocol
* No concurrent chronic systemic immune or hormone therapy, except neoadjuvant chemotherapy
* Absence of any severe organ insufficiency
* No pregnancy or breast feeding
* Written informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Active bacterial, viral or fungal infection
* Parenchymal liver disease (any stage cirrhosis)
* High risk of bleeding during biopsy (anticoagulants, esophageal varices)
* Esophageal squamous cell carcinoma
* Helicobacter pylori positive at the time of biopsy sampling
* Radiofrequency ablation of the oesophagus
* Psychiatric pathology capable of affecting comprehension and judgement faculty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with Barrett oesophagus or esophageal adenocarcinoma who meet the eligibility criteria are candidates for inclusion in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Identification of plasma biomarkers (micro RNAs) for early detection of esophageal adenocarcinoma | 4 years
  Identification of micro RNAs in plasma and tissue of patients with (non-)dysplastic Barrett's esophagus and EAC that are differentially abundant, compared to healthy plasma (healthy volunteers) or healthy tissue (patient-matched healthy esophagus biopsies).
Identification of plasma biomarkers (messenger RNAs) for early detection of esophageal adenocarcinoma | 4 years
  Identification of messenger RNAs in plasma and tissue of patients with (non-)dysplastic Barrett's esophagus and EAC that are differentially abundant, compared to healthy plasma (healthy volunteers) or healthy tissue (patient-matched healthy esophagus biopsies).
Identification of biomarkers (messenger RNAs) for therapy response prediction | 2 years
  Identification of a set of messenger RNAs that change during treatment (using longitudinally collected plasma samples) and that separate responders from non-responders to neo-adjuvant radiochemotherapy.

SECONDARY OUTCOMES:
Development of a quantitative Polymerase Chain Reaction (qPCR) test for clinical use | 1 year
  After development and validation on an independent cohort, this test should be evaluated in a second external cohort

CONTACTS AND LOCATIONS:
Overall Officials: Piet Pattyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University hospital Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No